CLINICAL TRIAL: NCT00325169
Title: A Randomised, Double-blind, Double Dummy, 3 Way Crossover Study Evaluating the Effects of a Combination of Seretide 50/500mcg Twice Daily Plus Tiotropium Bromide 18mcg Once Daily Compared With the Individual Agents (Tiotropium Bromide 18mcg Alone and Seretide50/500mcg Alone) in the Treatment of Subjects With COPD
Brief Title: SERETIDE Plus Tiotropium Versus Individual Components
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SCO104962
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Cross-over; Tiotropium; Triple; COPD; SERETIDE 50/500; Dyspnoea; Impulse oscillometry; Plethysmography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tiotropium + SERETIDE 50/500

SUMMARY:
This study was designed to evaluate the effects on lung function of a combination of SERETIDE 50/500mcg twice daily plus tiotropium bromide 18mcg once daily compared with the individual treatments (tiotropium bromide 18mcg once daily alone and SERETIDE 50/500mcg twice daily alone) in subjects with COPD. The study will utilise a three-way cross-over design with a 2-week wash-out period between each 2-week consecutive treatment period.

DETAILED DESCRIPTION:
A randomised, double-blind, double dummy, 3 way cross-over study evaluating the effects of SERETIDE™ 50/500mcg twice daily plus tiotropium bromide 18mcg once daily compared with the individual treatments (tiotropium bromide 18mcg alone and SERETIDE 50/500mcg alone) in the treatment of subjects with COPD

ELIGIBILITY:
Inclusion Criteria:

* Has an established clinical history of COPD as defined as per the GOLD definition.
* Post-bronchodilator FEV1 of >30% to 75% of predicted normal at Visit 1, a post-bronchodilator FEV1 / FVC ratio = 70%.
* Current or ex-smoker with a smoking history of > 10 pack-years.

Exclusion Criteria:

* Has unstable COPD (Chronic Obstructive Pulmonary Disease).
* Has a current medical diagnosis of asthma and/or allergic rhinitis or know respiratory disorders (lung cancer, sarcoidosis, tuberculosis or lung fibrosis) Requires regular (daily) or long term oxygen therapy (LTOT). (LTOT is defined as > 12 hours oxygen use per day).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-12; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
AUC (0-4hrs, sGAW after morning dose of medication at day 14)

SECONDARY OUTCOMES:
Effects of SERETIDE 50/500mcg twice daily plus tiotropium bromide 18mcg once daily compared with the individual treatments on further elements of lung function, dyspnoea, symptoms and a patient/physician assessment of treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Ghent, Belgium
- United Kingdom (3):
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Singh D, Brooks J, Hagan G, Cahn A, O'Connor BJ. Superiority of "triple" therapy with salmeterol/fluticasone propionate and tiotropium bromide versus individual components in moderate to severe COPD. Thorax. 2008 Jul;63(7):592-8. doi: 10.1136/thx.2007.087213. Epub 2008 Feb 1. PMID 18245142
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 104962 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104962 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104962 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104962 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104962 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104962 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104962 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register